CLINICAL TRIAL: NCT04359069
Title: Optimal Duration of Urinary Catheterization After Total Mesorectal Excision
Brief Title: Duration of Urinary Catheterization
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Sarah Koller, Assistant Professor of Clinical Surgery, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS-19-00633
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Surgery

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Non-inferiority Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urinary catheter removal on postoperative day 1 (Experimental)
  Interventions: Other: Urinary catheter removal on postoperative day 1
- Urinary catheter removal on postoperative day 3 (Active Comparator)
  Interventions: Other: Urinary catheter removal on postoperative day 3

INTERVENTIONS:
Other: Urinary catheter removal on postoperative day 1 — Urinary catheter will be removed on day 1 (experimental) instead of day 3 (standard of care).
  Arms: Urinary catheter removal on postoperative day 1
Other: Urinary catheter removal on postoperative day 3 — Urinary catheter will be removed on day 3 (standard of care)
  Arms: Urinary catheter removal on postoperative day 3

SUMMARY:
This study is being conducted to determine the length of time a urinary catheter is needed to drain urine from the bladder after colorectal surgery. Urinary retention is a well known complication after pelvic colorectal surgery, and current practice is to continue urinary catheterization for 3- days following pelvic colorectal surgery in an effort to avoid this complication. However, prolonged urinary catheterization is associated with increased risk of urinary tract infections as well as longer hospital stays. The investigators hypothesize that postoperative urinary catheters may be safely removed on postoperative day 1 without increased urinary retention rates. The purpose of this study is to evaluate whether a shorter duration of urinary catheterization (1 day) is non-inferior when compared to standard duration (3 days) in regards to postoperative urinary retention. The investigators plan to perform a prospective, randomized, non-inferiority trial comparing the urinary catheter duration of 1 day and 3 days with the primary endpoint of postoperative urinary retention. Secondary endpoints are urinary tract infection and length of hospital stay. The participants will be randomly assigned to the control group (catheter removal on postoperative day 3) or the experimental group (catheter removal on postoperative day 1).

DETAILED DESCRIPTION:
Disease Background:

Total mesorectal excision can be associated with transient post-operative urinary retention due to surgical disruption of pelvic autonomic nerves during procedure. These patients receive intra-operative urinary catheter to prevent post-operative urinary retention. However, the optimal duration for post-operative urinary catheter is not known, and longer duration of urinary catheter is associated with increased morbidity, such as urinary tract infection. A previous prospective randomized controlled trial from 1999 looking at this subject showed an increased rate of postoperative urinary retention in patients who had shorter duration of urinary catheterization. However, surgical techniques have improved significantly since then and a newer retrospective study comparing outcomes between patients who had catheter removal on postoperative day 1 vs catheter removal on day 2 or later demonstrated lower rates of urinary retention overall and there was no difference in rates of urinary retention between the two groups. A recent randomized non--inferiority trial investigating early urinary catheter removal in patients undergoing major colorectal surgery found that early removal, when combined with an oral alpha- antagonist, is non--inferior to standard removal and is associated with lower rates of urinary tract infections and shorter hospital stays.

Rationale:

A current prospective randomized trial is needed to determine the optimal duration of urinary catheterization in patients who receive total mesorectal excision (TME). Urinary catheterization is an established part of the intraoperative and postoperative care for this surgery. There should be minimal urinary dysfunction as total mesorectal excision should preserve pelvic autonomic nerve function with careful dissection. Current standard of practice is removal of urinary catheter on postoperative day 3. The study participants would be exposed to minimal risk as they would already require urinary catheterization as part of the standard of care. While this study will determine duration of postoperative urinary catheterization, it will not impact the surgical procedure itself. The control group would undergo removal of urinary catheter on postoperative day 3 and the experimental group would undergo removal of urinary catheter on postoperative day 1. The main risk endured by study participants would be the need to replace the urinary catheter if the patient has urinary retention following catheter removal. This study will contribute to existing knowledge by providing a prospective randomized non--inferiority trial investigating the impact of duration of urinary catheterization following total mesorectal excision on rates of postoperative urinary retention, urinary tract infections, and length of hospital stay. If shorter duration of urinary catheterization is shown to be non--inferior to standard duration of catheterization in terms of postoperative urinary retention, adopting a practice of catheter removal on postoperative day 1 may result in lower rates of catheter--associated urinary tract infections and shorter hospital stays. This practice would also adhere to the Surgical Care Improvement Project (SCIP) measures which recommend removal of urinary catheter on postoperative day 1 or 2. We hypothesize that postoperative urinary catheters may be safely removed on postoperative day 1 following total mesorectal excision without increased urinary retention rates when compared to removal on postoperative day 3.

Study Design:

This study will be conducted as a prospective, randomized, non-inferiority trial. The investigators will evaluate all patients undergoing total mesorectal excision for study eligibility. Consent for participation in the study will be obtained perioperatively. All male patients will be given a survey to assess their international prostate symptom severity (IPSS) score preoperatively. After surgery, the participant will be randomly assigned to the control (day 3 catheter removal) or experimental (day 1 catheter removal) group if there were no intraoperative complications deemed to interfere with the study, such as genitourinary tract injury requiring prolonged urinary catheterization postoperatively. Randomization will be performed using Microsoft Excel using a reported simple randomization method. The control group will have catheter removed at 9AM on postoperative day 3, while the experimental arm will have catheter removed at 9AM on postoperative day 1. Participants will receive appropriate maintenance IV fluids depending on their ability to tolerate PO intake postoperatively.

The primary endpoint of the study will be urinary retention, defined by grade 2 urinary retention per NCI CTCAE. Clinically, the investigators will identify these patients as those unable to void within 6 hours of urinary catheter removal with associated signs of suprapubic fullness and/or tenderness, and bedside ultrasound bladder scan showing more than 250cc of urine. Bladder scan will only be performed on patients who have signs of urinary retention and are unable to void within 6 hours of catheter removal. If subjects are unable to void spontaneously within 6 hours following catheter removal, a one-time straight catheterization will be performed, as per standard practice. If subjects are still unable to urinate within 6 hours following straight catheterization, an indwelling urinary catheter will be replaced. Secondary endpoints include urinary tract infection and length of hospital stay postoperatively. Urinary tract infection is defined as grade 2 or 3 urinary tract infection per NCI CTCAE. Patients will be evaluated for symptoms and signs of infection such as suprapubic pain, tenderness, dysuria, hematuria, and urinary frequency in addition to the presence of >100,000 colony-forming units/mL of bacteria on urine culture. Urinalysis and urine culture will only be sent in the setting of clinical signs and symptoms of urinary tract infection. Patients identified with UTI will be treated with pathogen-appropriate antibiotics as per standard practice. Length of hospital stay will be defined as the number of admitted days in the hospital from day of surgery to day of discharge. The participants will remain in the study until discharge from the hospital.

Data Collection:

Data regarding patient's demographic, past medical history, surgical indication, surgical approach, intraoperative complications, and postoperative outcomes including the mentioned endpoints will be collected prospectively through the electronic medical record system. The international prostate symptom severity (IPSS) score will be completed preoperatively for all male patients. Patient's medical record number will be numerically encoded and stored in a separate file. All paper documentation, including the original consent form, will be stored in a secure cabinet in the division office.

Follow up:

There will not be post-discharge follow up for the purpose of the research. Only data related to patient's history and inpatient hospital stay will be collected. Therefore, the follow up period for the endpoints is up to day of discharge.

Sample Size and Accrual:

Previous studies have identified rates of urinary retention following rectal surgery to approximately 20%. Given no expected difference between the two groups, the investigators therefore anticipate the urinary retention rate of both the study and control group to be 20%. Using a type I error of 5%, a power of 0.8, and a non-inferiority limit of 15% as reported by literature (3), a sample size of 88 per group will be needed. Given the anticipated rate of approximately 10 total mesorectal excision procedures per month, the investigators anticipate needing 18 months to fulfill the required sample size.

Data Analyses Plans:

The two randomized groups will be compared in terms of their preoperative demographics, prior history of benign prostatic hyperplasia, surgical indication, cancer staging, and neoadjuvant treatments. Intraoperative and postoperative factors will also be compared between the two groups. Subgroup analysis may be performed stratifying patients with different surgical indications and/or cancer staging. Given that the main research question involves patients following TME, regardless of surgical indication, the study may not be powered to observe differences when performing subgroup analyses.

Comparisons between groups will be analyzed by the chi square test, the Mann Whitney U test, or the Student t test for quantitative and qualitative variables, as appropriate. The early catheter removal will be considered noninferior to standard removal if the upper limit of a 1-sided 95% confidence interval excludes a difference in favor of the standard group of the standard group of more than 15%. A p-value of <.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Elective procedures involving total mesorectal excision, including low anterior resection and abdominoperineal resection for rectal cancer as well as proctectomy for inflammatory bowel disease.
* All approaches (open, laparoscopic and robotic) will be included, as the approaches not differ in the total mesorectal excision technique.
* Patients who received neoadjuvant chemotherapy and/or radiation treatments will be included.
* Age ≥ 18 years.
* American Society of Anesthesiologists (ASA) class I-III.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Patients undergoing emergent or urgent surgery.
* Patients undergoing total mesorectal excision in combination with other major surgical procedures on the same day should be excluded from this study.
* Patients sustaining genitourinary tract injury during the procedure should be excluded postoperatively.
* History of urinary retention after previous procedure, surgery, or urinary catheter removal.
* History of urinary retention not being actively treated.
* Patients requiring prolonged duration or replacement of urinary catheter in the postoperative period for reasons other than urinary retention should be excluded.
* History of neurogenic bladder.
* Patients with chronic indwelling Foley catheterization or suprapubic catheterization.
* History of cystectomy and/or any surgically created urinary conduit, including neobladder and ileal conduit.
* Patients less than 18 years of age should be excluded from this study.
* Vulnerable patients including incarcerated patients or any patients unable or unwilling to provide informed consent will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Rate of urinary retention | From time of surgery to time of discharge from the hospital, an average of 4 days

SECONDARY OUTCOMES:
Rate of urinary tract infection | From time of surgery to time of discharge from the hospital, an average of 4 days
Length of hospital stay | From time of surgery to time of discharge from the hospital, an average of 4 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Keck Hospital of USC, Los Angeles, California
  - Los Angeles County Hospital (LAC/USC), Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benoist S, Panis Y, Denet C, Mauvais F, Mariani P, Valleur P. Optimal duration of urinary drainage after rectal resection: a randomized controlled trial. Surgery. 1999 Feb;125(2):135-41. PMID 10026745
- [Background] Yoo BE, Kye BH, Kim HJ, Kim G, Kim JG, Cho HM. Early Removal of the Urinary Catheter After Total or Tumor-Specific Mesorectal Excision for Rectal Cancer Is Safe. Dis Colon Rectum. 2015 Jul;58(7):686-91. doi: 10.1097/DCR.0000000000000386. PMID 26200683
- [Background] Patel DN, Felder SI, Luu M, Daskivich TJ, N Zaghiyan K, Fleshner P. Early Urinary Catheter Removal Following Pelvic Colorectal Surgery: A Prospective, Randomized, Noninferiority Trial. Dis Colon Rectum. 2018 Oct;61(10):1180-1186. doi: 10.1097/DCR.0000000000001206. PMID 30192326
- [Background] Kwaan MR, Lee JT, Rothenberger DA, Melton GB, Madoff RD. Early removal of urinary catheters after rectal surgery is associated with increased urinary retention. Dis Colon Rectum. 2015 Apr;58(4):401-5. doi: 10.1097/DCR.0000000000000317. PMID 25751796
- [Background] Kin C, Rhoads KF, Jalali M, Shelton AA, Welton ML. Predictors of postoperative urinary retention after colorectal surgery. Dis Colon Rectum. 2013 Jun;56(6):738-46. doi: 10.1097/DCR.0b013e318280aad5. PMID 23652748
- [Background] Kim J, Shin W. How to do random allocation (randomization). Clin Orthop Surg. 2014 Mar;6(1):103-9. doi: 10.4055/cios.2014.6.1.103. Epub 2014 Feb 14. PMID 24605197
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542